CLINICAL TRIAL: NCT01460303
Title: Clinical Trial of Patient Operated Valved Catheter Compared With Standard Indwelling Transurethral Catheter for Postoperative Bladder Management
Brief Title: Patient-operated Valved Catheter Versus Indwelling Transurethral Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Michael Flynn, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-13523
Record Dates: First submitted 2011-10-19; First posted 2011-10-26 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Bladder Dysfunction; Urinary Retention
Keywords: Transurethral catheterization; Urinary retention; Bladder dysfunction; Patient comfort; Pelvic Reconstructive Surgery; Postoperative bladder dysfunction; Postoperative urinary retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPTION-vf patient controlled catheter (Experimental): Patients who fail postop bladder challenge and are randomized to "OPTION-vf" arm will be instructed in the use and care of this catheter, discharged home with it in place and given an appointment between 5-10 days postop for a bladder challenge.
  Interventions: Device: Bladder catheter: OPTION-vf patient controlled catheter vs. indwelling transurethral catheter with leg bag
- Transurethral catheter w/leg bag (Active Comparator): Patients who fail postop bladder challenge and are randomized to "indwelling catheter with leg bag" arm will be instructed in the use and care of this catheter, discharged home with it in place and given an appointment between 5-10 days postop for a bladder challenge.
  Interventions: Device: Transurethral catheter with leg bag

INTERVENTIONS:
Device: Bladder catheter: OPTION-vf patient controlled catheter vs. indwelling transurethral catheter with leg bag — OPTION-vf patient controlled catheter (transurethral catheter with external drainage valve to provide on-demand drainage of urine stored directly from the bladder), worn maximum of 30 days post-op until bladder challenge is passed. Bladder challenge is considered "passed" when a patient is able to void adequately and spontaneously (without the assistance of a catheter).
  Other Names: OPTION-vf™ Valved Female Urinary Catheter; Patient Controlled Catheter
  Arms: OPTION-vf patient controlled catheter
Device: Transurethral catheter with leg bag — Transurethral catheter w/leg bag urine storage, worn maximum of 30 days post-up until bladder challenge is passed. Bladder challenge is considered "passed" when a patient is able to void adequately and spontaneously (without the assistance of a catheter).
  Other Names: Foley catheter
  Arms: Transurethral catheter w/leg bag

SUMMARY:
Following surgery for female urinary incontinence and/or pelvic organ prolapse, women are sometimes temporarily unable to empty their bladders and are sent home with a transurethral indwelling catheter attached to a bag which holds urine. The goal of this study is to compare a new type of patient-operated catheter without a bag to the catheter with a bag for ease of use, comfort and quality of life for patients during the postoperative recovery period. This new catheter, the OPTION-vf, is approved by the FDA and is available on the market.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery for urinary incontinence and/or pelvic organ prolapse at the UMass Memorial Medical Center with one of the Urogynecology/Reconstructive Pelvic Surgery faculty.

Exclusion Criteria:

* inability to provide consent
* <18 years old
* non-English speaking
* patients using intermittent self-catheterization
* patients sustaining bladder injury during surgery
* prisoners
* pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Flynn, MD, Principal Investigator — University of Massachusetts, Worcester

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OPTION-vf Patient Controlled Catheter | Transurethral Catheter w/Leg Bag
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPTION-vf Patient Controlled Catheter | Transurethral Catheter w/Leg Bag | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (12.4) | 59.7 (12.4) | 60.6 (1.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 21 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Total Catheter Related Pain
Description: Total Catheter Related Pain Range Scale (0 = none, to 10 = worst) on the Post Operative Questionnaire All subjects were given and appointment for an outpatient voiding trial after hospital discharge. The Post Operative questionnaire was completed by the subject one time at that appointment.
Time Frame: 5-10 days postoperatively
Measure: Median (Standard Deviation); unit: units on a scale
Groups:
- OPTION-vf Patient Controlled Catheter: Patients who fail postop bladder challenge and are randomized to "OPTION-vf" arm.
  Bladder catheter: OPTION-vf patient controlled catheter vs. indwelling transurethral catheter with leg bag: OPTION-vf patient controlled catheter (transurethral catheter with external drainage valve to provide on-demand drainage of urine stored directly from the bladder), worn maximum of 30 days post-op until bladder challenge is passed. Bladder challenge is considered "passed" when a patient is able to void adequately and spontaneously (without the assistance of a catheter).
- Transurethral Catheter w/Leg Bag: Patients who fail postop bladder challenge and are randomized to "indwelling catheter with leg bag" arm.
  Transurethral catheter with leg bag: Transurethral catheter w/leg bag urine storage, worn maximum of 30 days post-up until bladder challenge is passed. Bladder challenge is considered "passed" when a patient is able to void adequately and spontaneously (without the assistance of a catheter).
Arm/Group | OPTION-vf Patient Controlled Catheter | Transurethral Catheter w/Leg Bag
Number analyzed (Participants) | 24 | 25
units on a scale | 1.25 (2.65) | 2.3 (3.5)

2. Secondary Outcome: Composite Satisfaction Score (CSS)
Description: The mean scores for the first 5 questions of the Post Operative Questionnaire were used to calculate a Composite Satisfaction Score.
  1. Total Pain (0 none, 10 worst)
  2. Total Catheter Related Pain Range Scale (0 none, 10 worst)
  3. Ease of catheter use (0 easy, 10 difficult)
  4. Feeling of frustration (0 none, 10 very much)
  5. Limited social activities (0 none, 10 very much) All subjects were given and appointment for an outpatient voiding trial after hospital discharge. The Post Operative Questionnaire was completed by the subject one time at that appointment.
Time Frame: 5-10 days postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OPTION-vf Patient Controlled Catheter | Transurethral Catheter w/Leg Bag
Number analyzed (Participants) | 24 | 25
units on a scale | 2.23 (1.83) | 3.62 (1.95)

ADVERSE EVENTS:
Time Frame: Up to six weeks after placement of catheter
Arm/Group | OPTION-vf Patient Controlled Catheter | Transurethral Catheter w/Leg Bag
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 11/24 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPTION-vf Patient Controlled Catheter (N=24) | Transurethral Catheter w/Leg Bag (N=25)
Urinary Tract Infection (Renal and urinary disorders) | 11 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes